CLINICAL TRIAL: NCT02390518
Title: Phase I Study of Stereotactic Radiosurgery Dose Escalation for Brain Metastases
Brief Title: Stereotactic Radiosurgery Dose Escalation for Brain Metastases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI71940
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Stereotactic Radiosurgery (Experimental)
  Interventions: Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery — Patients with 1 to 5 brain metastases will be treated. Patients will be assigned to one of four cohorts based on the size of their brain lesions. For each patient, a single lesion will be treated at experimental dose level, other metastases (if present) will receive standard SRS doses.
  Dose Level 1 Dose Level 2 Dose Level 3 Dose Level 4 Cohort 1a and 1a Expansion (starting at Dose Level 3) Diameter: ≤ 10 mm Volume: ≤ 0.5236 cm3 26 Gy 28 Gy 30 Gy n/a Cohort 1b Diameter: 11-20 mm Volume: 0.5237-4.1888 cm3 26 Gy 28 Gy 30 Gy n/a *Cohort 2 Diameter: 21-30 mm Volume: 4.1889-14.1372 cm3 20 Gy 22 Gy 24 Gy n/a
  **Cohort 3 Diameter: 31-40 mm Volume: 14.1373-33.5103 cm3 17 Gy 19 Gy 21 Gy 23 Gy
  Dose Escalation A non-standard 5+4 design will be used for the dose escalation. For each cohort, an initial group of 5 patients will be accrued at dose level 1 and receive experimental treatment to one of their lesions.
  Other Names: SRS

SUMMARY:
This is a Phase I dose escalation and expansion trial. The purpose of this study is to determine the maximum tolerated dose of radiation received during stereotactic radiosurgery in patients with brain metastases who have never received radiation to the brain before.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed brain metastases by CT or MRI criteria. If there is evidence of extra-cranial metastatic disease, it is preferable that the lesions be pathologically confirmed (see section 4.2.5 for excluded histologies) and reviewed by a University of Utah or Huntsman Cancer Hospital pathologist if the initial review was done at an outside facility.
* Prior brain surgery is allowed, although a lesion situated in the operative bed would not be selected to receive an experimental dose of SRS treatment. SRS should be delivered 4-6 weeks post-surgery if the patient had a craniotomy for resection of a lesion. Enrollment of a patient with the goal of performing SRS outside of the 4-6 post-craniotomy window is at the PI's discretion.
* Patients must have 1-5 untreated brain metastases total.
* For patients planning to enroll in Cohort 1a (including expansion) or Cohort 1b: Tumor volume ≤ 4.1888 cm3 by CT or MRI measurement at the time of consultation/screening for the metastatic lesion on trial. Patients who have at least one additional lesion that is larger than the lesions eligible for the expansion cohort, but who are unable to find another open cohort, will have the eligible lesion(s) treated in the expansion cohort, and the remaining lesion(s) treated at the standard dose.

For patients enrolling in the expansion Cohort 1a: Up to five brain metastases with tumor volume ≤ 0.5237 cm3 by CT or MRI measurement at the time of consultation/screening will be treated on trial with the MTD. Brain metastases with volume > 0.5237 cm3 will be treated by standard of care SRS dosing.

For patients enrolling in Cohort 1b: Tumor volume of > 0.5237 cm3 and ≤ 4.1888 cm3 by CT or MRI measurement at the time of consultation/screening for the metastatic lesion on trial. All other brain metastases will be treated by standard of care SRS dosing.

* As of Protocol Version 9, Cohorts 2 and 3 are permanently closed to accrual. For patients planning to enroll in Cohort 2 or 3: Equivalent tumor diameter ≤ 40 mm by CT or MRI measurement at the time of consultation/screening for the metastatic lesion on trial. Equivalent tumor diameter </=40 mm by CT or MRI measurement for all lesions treated by standard of care SRS dosing.
* All metastatic lesions must be separated by a minimum of 3 cm as measured from the peripheral edges of the lesions that are in closest proximity to one another. If multiple lesions are present and are not all ≥ 3 cm away from each other, the patient will be deemed ineligible.
* Prior systemic therapy is allowed, although appropriate washout is required for patients who have been on BRAF inhibitors (at least 7 days).
* For subjects currently on active systemic cancer therapy, the treating medical oncologist should be consulted to ensure proper washout (if appropriate) periods prior to SRS.
* Patients must be at least 18 years of age.
* Karnofsky Performance Status (KPS) ≥ 60.
* Able to provide informed consent and have signed an approved consent form that conforms to federal and institutional guidelines.
* Women of child-bearing potential must have a negative pregnancy test within 10 days of study enrollment and must agree to use an acceptable method of birth control while receiving radiation and for 3 months after radiation. Women of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for >1 year.
* Men who are able to father a child must agree to use an acceptable method of birth control while receiving radiation, and for 3 months after radiation.

Exclusion Criteria:

* Prior whole/partial brain irradiation.
* Brain lesions with an equivalent diameter of > 40 mm in size on MRI imaging at the time of consultation/screening for protocol eligibility.
* Lesions located in anatomic regions that are not amendable to SRS (e.g., optic nerve)
* Brain lesions located in the brain stem.
* Radiographic or cytologic evidence of leptomeningeal disease
* Primary lesion with radiosensitive histology that includes the following: small cell carcinoma, germ cell tumors, lymphoma, leukemia, or multiple myeloma
* Women of child-bearing potential who are pregnant or breast feeding
* Patients with multiple lesions, which by size criteria would be enrolled in a cohort which is full at the time of enrollment and the 12 weeks DLT period has not been reached.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-05-07 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of stereotactic radiosurgery | Maximum Tolerated Dose of stereotactic radiosurgery will be evaluated throughout the treatment period which is expected to last 12 weeks per patient
  Patients will be evaluated for any grade 3 or greater toxicities attributed to the lesion treated with the escalated dose

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No